CLINICAL TRIAL: NCT06730009
Title: A Dose-Finding Phase I Followed by a Phase II Study to Evaluate the Safety and Efficacy of Allogeneic NK-cell Combined With Chemotherapy in Patients With PDA or Cholangiocarcinoma After Surgery
Brief Title: Phase I/II Study: Allogeneic NK-cell Therapy With Chemotherapy for Post-Surgery PDA or Cholangiocarcinoma Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-ANK-21
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Carcinoma Stage II; Cholangiocarcinoma Resectable
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLOG + Allogeneic NK cells (Experimental): Ph I SLOG + Allogeneic NK cell dose escalation (Cohort 1:10 × 10^8 cells ; Cohort 2:20 × 10^8 cells) Ph II Arm 1 SLOG + Allogeneic NK cell
  Interventions: Biological: SLOG + Allogeneic NK cell
- SLOG chemotherapy (Active Comparator): Ph II Arm 2
  Interventions: Drug: SLOG chemotherapy

INTERVENTIONS:
Biological: SLOG + Allogeneic NK cell — Drug: SLOG chemotherapy S-1, leucovorin, oxaliplatin, and gemcitabine (SLOG)
  Biological:
  Allogeneic Magicell-NK contains NK cells suspended in 100 mL of normal saline Ph I dose starts at 10 × 10^8 cells (Cohort 1) and escalates to 20 × 10^8 cells (Cohort 2).
  Ph II dose will be determined lower than or equal to Ph I MTD/MFD.
  Arms: SLOG + Allogeneic NK cells
Drug: SLOG chemotherapy — Drug: SLOG chemotherapy S-1, leucovorin, oxaliplatin, and gemcitabine (SLOG)
  Arms: SLOG chemotherapy

SUMMARY:
This is a phase I/II study which intends to characterize the safety, tolerability, and preliminary efficacy of Allogeneic Magicell-NK infusion in PDA or cholangiocarcinoma patients after surgery. Subjects will receive a total of 6 intravenous (IV) infusions of the IP on the 11th day of each chemotherapy cycle. A total of 6 cycles of IP infusions are planned.

The phase I part of the study is a first-in-human phase I trial of Allogeneic Magicell-NK and is therefore designed in an open-label, dose-escalation manner. A standard 3+3 design will be employed to assess the safety profile of Allogeneic Magicell-NK and to determine the MTD/MFD. Two dose cohorts are planned: the starting dose is 10 × 10^8 cells (Cohort 1), and escalates to 20 × 10^8 cells (Cohort 2).

The phase II part of the study is designed as an open-label, two-arm, randomized clinical trial comparing the combination of SLOG and Allogeneic Magicell-NK with SLOG alone when used as adjuvant therapy following resection for PDA or Cholangiocarcinoma. Approximately 30 subjects will be randomized at a 2:1 ratio between the two arms: Arm 1: SLOG and Allogeneic Magicell-NK (20 subjects); Arm 2: SLOG alone (10 subjects). Subjects will then receive 12 weeks of SLOG chemotherapy with or without Allogeneic Magicell-NK infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Dated and signed informed consent.
2. Either sex, aged older than 18 years old (inclusive) at date of consent.
3. Subject with a macroscopic resection of the primary tumor and residual primary tumor that satisfies all of the items below according to the Union for International Cancer Control (UICC) histopathologic staging system:

   * At or before the surgery, stage II or stage III.
   * Local residual tumor classified as R0 or R1.
   * Cytologic examination negative upon intraoperative peritoneal lavage.
4. Histologically confirmed PDA or cholangiocarcinoma.
5. Received curative resection within 12 weeks prior to screening visit and will receive adjuvant SLOG chemotherapy. Note: Subjects with cancer who had undergone surgery with or without prior neo-adjuvant therapy will be recruited.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
7. Subject with adequate hematology function at Visit 1:

   * Total white blood cell (WBC) ≥ 3,000 cells/mm3.
   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3.
   * Platelets ≥ 100,000 counts/mm3.
   * Hemoglobin ≥ 9 g/dL.
   * International normalized ratio (INR) of prothrombin time within normal range. Note: Re-test for eligibility is allowed during the screening period.
8. Subject with adequate hepatic and renal function at Visit 1:

   * Serum creatinine ≤ 1.5× Upper Limit of Normal (ULN).
   * Blood urea nitrogen (BUN) ≤ 1.5× ULN.
   * Total bilirubin ≤ 1.5× ULN.
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5× ULN.
   * Alkaline phosphatase (ALP) ≤ 5× ULN.
   * Albumin ≥ 3.0 g/dL. Note: Re-test for eligibility is allowed during the screening period.
9. Negative response in human immunodeficiency virus (HIV) and treponema pallidum (rapid plasma reagin [RPR]/venereal disease research laboratory [VDRL] and treponema pallidum hemagglutination [TPHA]).
10. Subject confirmed with past cytomegalovirus (CMV) infection in terms of having positive CMV immunoglobin G (CMV IgG).
11. Subject with childbearing potential must agree to use at least two contraceptive precautions, one of which must be a condom or other adequate barrier method, from

    * signing informed consent until 28 days after the last dose of investigational product (IP) administration.
    * initiation of oxaliplatin treatment until at least 15 months (female) or 12 months (male) following the last dose.
    * initiation of gemcitabine treatment until at least 6 months (female) or 3 months (male) following the last dose.
12. Agree to be in compliance with clinical protocol-planned treatment. Note: Anti-virus treatment is allowed if active hepatitis B is presented.

Exclusion Criteria:

1. Received any other investigational, anti-neoplastic medications, or immune cell therapy within 28 days prior to screening visit.
2. Any prior history of malignant neoplasm, except:

   1. Non-invasive, non-melanomatous skin cancer (including squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ), curatively treated with cryosurgery or surgical excision only.
   2. Other primary malignant neoplasm diagnosed as disease free for more than 5 years.
3. Immunocompromized, currently under immunosuppressive treatment for autoimmune disease, or have received systemic steroid of equivalent dosage higher than prednisolone 30 mg/day for more than 7 days within 14 days prior to Day 1.
4. With known metastases.
5. With ongoing acute diseases, or serious medical conditions within the past 2 years prior to screening, such as cardiovascular (e.g., New York Heart Association grade III or IV), hepatic (e.g., Child-Pugh Class C), psychiatric condition (e.g., alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject.
6. Hypercoagulable state that may lead to clinically apparent thrombosis.
7. With known hypersensitivity to aminoglycoside (e.g., streptomycin, gentamicin) or bacitracin.
8. With known hypersensitivity to any of the components of Allogeneic Magicell-NK, including human serum albumin.
9. With known hypersensitivity to any of the components of S-1, leucovorin, oxaliplatin, or gemcitabine.
10. With any contraindication to S-1, leucovorin, oxaliplatin, or gemcitabine, including:

    - Severe myelosuppression or myelosuppression that probably exacerbates.
11. With symptomatic CMV disease.
12. With any history of diagnosed or suspected cardiac arrhythmia or QT interval prolongation.
13. Male subject with a corrected QT interval (QTc) ≥ 450 ms and female subject with a QTc ≥ 470 ms as determined by electrocardiogram (ECG) examination at screening.
14. Received any drugs associated with QT prolongation within 28 days prior to the Screening Visit (refer to Appendix 3. Drugs Associated with QT Prolongation, including but not limited to the drug listed therein).
15. Received brivudine or its analogs (e.g., sorivudine) or any live vaccines within 28 days prior to the Screening Visit.
16. Female subject who is lactating or has positive serum or urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Ph I Evaluation of safety parameters, numbers of participants with Treatment-Emergent Adverse Events (TEAEs). | 15 months
  The number of participants with Treatment-Emergent Adverse Events (TEAEs) was assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) to assess the tolerability of Magicell-NK treatment.
Ph I Laboratory tests | 15 months
  Number of participants with abnormal laboratory test results.
Ph I Body weight | 5 months
  Body weight (KG) will be measured at baseline, treatment, and F1 visits. The number of participants with abnormal body weight change.
Ph I Vital signs | 15 months
  Number of participants with abnormal vital signs.
Ph I Dose-limiting toxicities | 4 months
  Adverse events were assessed according to NCI-CTCAE v5.0 criteria.
Ph I Maximum Tolerated Dose (MTD) and Recommended Phase II Dose | 4 months
  MTD is defined as the highest dose level at which ≤ 1/6 of subjects experienced DLT.
Ph II Disease-free survival (DFS) | 15 months
  The time from the date of the first Magicell-NK infusion to the date of the first disease-free survival event (recurrence, second primary PDA or Cholangiocarcinoma, or death from any cause).

SECONDARY OUTCOMES:
Ph I Disease-free survival (DFS) | 15 months
  The time from the date of the first Magicell-NK infusion to the date of the first disease-free survival event (recurrence, second primary PDA or Cholangiocarcinoma, or death from any cause)
Ph II Evaluation of safety parameters, numbers of participants with Treatment-Emergent Adverse Events (TEAEs) | 15 months
  The number of participants with Treatment-Emergent Adverse Events (TEAEs) was assessed using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) to assess the tolerability of Magicell-NK treatment.
Ph II Laboratory tests | 15 months
  Number of participants with abnormal laboratory test results.
Ph II Body weight | 5 months
  Body weight (KG) will be measured at baseline, treatment, and F1 visits. The number of participants with abnormal body weight change.
Ph II Vital signs | 15 months
  Number of participants with abnormal vital signs.
Ph I/II Tumor recurrence rate (TRR) | 15 months
  To evaluate the Tumor recurrence rate (TRR) during the study period
Ph I/II Changes in Frequency and Duration of ctDNA | Up to 15 months
  Number of participants experiencing ctDNA seroconversion (i.e. ctDNA+ that become ctDNA-) after any Allogeneic Magicell-NK regimen remaining disease free
Ph I/II Changes in Frequency and Duration of Circulating Tumor Count (CTC) | Up to 15 months
  Determine the effect of Allogeneic Magicell-NK on reducing CTC of whole blood in the subject with elevated baseline CTC count to identify the least effective dose that clears CTCs. The baseline count of CTC will be recorded before Allogeneic Magicell-NK therapy in a whole blood sample. In the treatment, the count of CTC will be measured at C4D1 and each follow-up visit after Allogeneic Magicell-NK therapy in a whole blood sample. All of these values will be compared.
Ph I/II Changes in Biomarkers (CA19-9 and CEA) | Up to 15 months
  Determine the effect of Allogeneic Magicell-NK on CEA and CA 19-9 in the subject with elevated baseline CEA and CA 19-9 to identify the least effective dose that clears CEA and CA 19-9. The baseline count of CEA and CA 19-9 will be recorded before Allogeneic Magicell-NK therapy. In the treatment, the count of CEA and CA 19-9 will be measured at C4D1. And each follow-up visit after Allogeneic Magicell-NK therapy. All of these values will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Chang, PhD, Study Chair — Medigen Biotechnology Corporation
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No